CLINICAL TRIAL: NCT05828108
Title: A Phase I/II, Intra-Patient Dose-Escalation Study of the Selective GlyT1 Inhibitor, Bitopertin for Steroid-Refractory Diamond-Blackfan Anemia.
Brief Title: Study of the Selective GlyT1 Inhibitor Bitopertin for Steroid-Refractory Diamond-Blackfan Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001528; 001528-H
Record Dates: First submitted 2023-04-22; First posted 2023-04-25 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09-16

CONDITIONS: Steroid-refractory Diamond-Blackfan Anemia (DBA)
Keywords: Inherited Bone Marrow Failure Syndrome; Erythroid Aplasia; Iron Homeostasis; Ribosomopathy; Heme Synthesis; Hemoglobin Synthesis
MeSH Terms: conditions — Congenital Bone Marrow Failure Syndromes; Anemia, Aplastic | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental -Bitopertin (Experimental): Bitopertin, up to a maximum dose of 60 mg (5 mg, 10mg, 20mg, 40mg, 60mg)
  Interventions: Drug: Bitopertin

INTERVENTIONS:
Drug: Bitopertin — Dose Escalation: Monthly (every 4 weeks) up to a maximum dose of 60 mg bitopertin (5 mg, 10mg, 20mg, 40mg, 60mg). At each monthly (4 week) interval, a complete blood count (CBC) with differential and a reticulocyte analysis (including reticulocyte hemoglobin) will be collected prior to taking the higher dose. If the absolute reticulocyte count (ARC) is 60,000 /microL or higher, the subject will hold at the current dose level (or return to that level if escalation has already occurred) for an additional 4 weeks. If, after 8 weeks at that dose, response criteria are met this will be considered the minimum effective dose (MED) and shall be the treatment dose throughout the remainder of the study unless modifications are indicated.

SUMMARY:
Background:

Diamond-Blackfan anemia (DBA) is an inherited disease that affects the bone marrow. People with DBA have chronic anemia that can be severe. Many must have frequent transfusions of red blood cells. Current treatments for DBA all have risks of serious side effects. Better treatments are needed.

Objective:

To test a new drug (bitopertin) in people with DBA.

Eligibility:

People aged 18 or older with DBA.

Design:

Participants will be screened. They will have a physical exam; they will have blood tests and a test of their heart function. They will have a bone marrow biopsy: An area of their hip will be numbed, and a needle will be inserted to remove a sample of tissue from inside the bone.

Bitopertin is a pill taken by mouth. Participants will take the drug once a day every day for 8 months. They will start with a low dose of the drug; the dosage may increase gradually over time. They will keep a diary to record each dose.

Participants will have blood tests every 4 weeks. This may be done in the clinic. Participants may also have telehealth visits; they can have blood drawn at a local lab and sent to the researchers.

The bone marrow biopsy and other tests will be repeated after 8 months.

Participants who have a positive response to bitopertin will be invited to enter an extended phase of the trial. They may continue to take the drug for 3 more years.

Those who choose not to continue in the extended phase may have a follow-up visit 6 months after they stop taking the drug.

DETAILED DESCRIPTION:
Study Description:

Diamond-Blackfan anemia (DBA) is an inherited bone marrow failure syndrome characterized by selective erythroid defects. In DBA, a defect in erythroid ribosome biosynthesis creates an asynchrony between protein synthesis of globin chains and heme, wherein the continued production of free heme without sufficient globin is toxic to cells. Bitopertin prevents the uptake of glycine through the GlyT1 transporter reducing the synthesis of 5- aminolevulinic acid, the rate-limiting step in heme synthesis, which in turn leads to a significant reduction in intracellular heme.

We hypothesize that bitopertin will rescue DBA by rebalancing heme and globin chain production and reducing the toxicity to the hematopoietic cells that the excess heme causes. Thus, we propose a phase I/II (pilot), single-arm, intra-patient dose-escalation trial of bitopertin for the treatment of steroid-refractory DBA.

Objectives:

Primary Objective: Efficacy of bitopertin in treating Diamond- Blackfan anemia

Secondary Objectives:

* Examine the safety and tolerability of bitopertin in treating Diamond-Blackfan anemia.
* Examine the maintenance of response and relapse rates of Diamond-Blackfan anemia during long-term bitopertin use
* Examine the effects of long-term treatment of Diamond-Blackfan anemia with bitopertin on clonal evolution, survival, and health- related quality of life metrics

Tertiary/Exploratory Objectives:

* Evaluate the impact of bitopertin on stem cell and erythroid cell dynamics in the Diamond-Blackfan anemia through correlative and translational studies
* Examine the pharmacology of bitopertin in Diamond-Blackfan anemia

Endpoints:

Primary endpoint:

-response rate from drug initiation until 8 months (32 weeks) as measured by an increase in pre-transfusion hemoglobin and/or either decrease in transfusion rate or transfusion-independence

Secondary endpoints:

* toxicity profile at 8 months (CTCAE criteria)
* intra-patient maximum tolerated dose at 8 months (32 weeks) from drug initiation
* response rate after 3 months (12 weeks) at the maximum tolerated dose
* response rate 3 years post-primary endpoint (extension)
* rate of relapse ongoing for up to 3 years, beginning 8 months (32 weeks) from drug initiation as demonstrated by new or increasing transfusion requirements and/or according to clinical outcome
* rate of clonal evolution on bitopertin annually for up to 3 years, beginning 8 months (32 weeks) from drug initiation as measured by karyotypic, histologic, and flow cytometric changes
* rate of overall survival ongoing for up to 3 years, beginning 8 months (32 weeks) from drug initiation according to clinical outcomes
* Health-related quality of life (HRQL) annually for up to 3 years, beginning 8 months (32 weeks) from drug initiation based on questionnaire-based inventory of HRQL

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Diamond-Blackfan anemia defined as chronic anemia presenting on or before the third year of life, associated with reticulocytopenia and greatly reduced or absent bone marrow erythroid precursors, supported by, but not requiring either:

   1. familial history
   2. gene mutation testing demonstrating a known disease-causing mutation or a mutation of disease-associated gene in combination with clinical characteristics of DBA

   Patients with late-onset DBA (diagnosed after the third year of life) may also be included if (but only if) gene mutation testing confirms a disease-causing mutation, as above.
2. Clinically-significant anemia as defined as either:

   1. hemoglobin less than 9.0 g/dL
   2. red cell transfusion of at least 2 units PRBC for adults in the eight weeks prior to study enrollment
3. Relapsed and/or steroid-refractory disease or patient intolerance of systemic corticosteroids
4. Age >= 18 years at the time of consent

Although all patients without a molecular diagnosis (i.e., genetic testing positive for a disease- causing lesion) will undergo targeted gene panel testing for mutations in all known genes associated with DBA , the diagnosis of DBA is a clinical one, and as such, consent and enrollment does not require results from these genetic tests in the absence of any features that would suggest an alternative diagnosis (e.g., Fanconi Anemia, Dyskeratosis Congenita, etc.).

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Treatment with androgens (danazol or oxymetholone) or corticosteroids less than 4 weeks prior to initiating bitopertin.

   -Stable physiologic dose steroid replacement for adrenal insufficiency or other similar conditions is not an exclusion criterium.
2. Hypersensitivity to bitopertin or its components
3. Patient Health Questionnaire-8 (PHQ-8) score greater than or equal to 10 or imminent suicidal risk identified by the Columbia-Suicide Severity Rating Scale (C-SSRS) as defined as suicidal ideation with intent (grade 4 or 5) within the last year or any suicidal behavior within the last five years
4. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy
5. Life expectancy of less than 3 months from any cause
6. History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

   * Recent myocardial infarction (within last 6 months),
   * Uncontrolled congestive heart failure,
   * Unstable angina (within last 6 months),
   * Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third-degree AV block without a pacemaker.)
   * Long QT syndrome, family history of idiopathic sudden death, congenital long QT syndrome or additional risk factors for cardiac repolarization abnormality, as determined by the investigator
   * Impaired cardiac function such as corrected QTc>450msec using Fridericia correction on the screening ECG, other clinically significant cardio-vascular disease (e.g., uncontrolled hypertension, history of labile hypertension), history of known structural abnormalities (e.g. cardiomyopathy).
7. Known active or uncontrolled infections not adequately responding to appropriate therapy.

   * Note, HIV infection is not exclusive of trial participation if the infection is effectively controlled with medications not known to interfere with bitopertin metabolism or be metabolized by pathways known to be altered by bitopertin. HIV RNA viral load must be undetectable at the time of enrollment, and CD4 cell count must be >= 200/microL. Patients must remain on antiretroviral therapy throughout study participation and must be periodically monitored for suppression of viral load and CD4 cell count.
   * If drug-drug interactions between antiretroviral (e.g. HIV), antiviral (e.g., hepatitis), or antifungal medications and bitopertin are suspected (such as lopinavir, ritonavir or other strong CYP3A4 inhibitors), these must be addressed by a qualified clinical pharmacist or pharmacologist, and any changes to antiretroviral therapy need to be approved in consultation with an Infectious Disease and/or HIV specialist prior to enrollment.
8. Evidence for MDS or AML as defined by WHO criteria, or any active malignancy or likelihood of recurrence of malignancies within 12 months
9. Patients who have received chemotherapeutic treatment or other specific antineoplastic drugs or radiation therapy within 6 months of study entry
10. Female subjects who are nursing or pregnant (positive serum or urine beta-human chorionic gonadotrophin (beta-hCG) pregnancy test) at screening/baseline visit
11. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, not using highly effective methods of contraception during dosing and for 30 days after the last dose of bitopertin. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post- ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate

    <1%), for example hormone vaginal ring or transdermal hormone contraception.
    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

      -Women are considered post-menopausal and not of childbearing potential if they have had over 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile age appropriate (e.g., generally 40-59 years), history of vasomotor symptoms (e.g., hot flushes) in the absence of other medical justification or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment should she be considered not of childbearing potential.
    * Sexually active males unless they use a condom during intercourse while taking the study treatment and for 30 days after stopping study treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via seminal fluid.
12. Active alcohol/drug abuse.
13. Unable to understand the investigational nature of the study or give informed consent and does not have a legally authorized representative or surrogate that can provide informed consent.
14. Unable to take the oral study drug.
15. Concurrent participation in an investigational study within 30 days prior to enrollment or within 5-half-lives of the study drug, whichever is longer. Note: parallel enrollment in a disease registry is permitted.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Rate of response | On a rolling basis (sliding window) from drug initiation until 8 months (32 weeks)
  Response as demonstrated by either an increase in hemoglobin or decrease in transfusion rate, and robust response as demonstrated by transfusion independence.

SECONDARY OUTCOMES:
Rate of relapse | Ongoing for up to 3 years, beginning 8 months (32 weeks) from drug initiation
  Relapse as demonstrated by new or increasing transfusion requirements and/or according to clinical outcome
Long-term safety of drug | Ongoing for up to 3 years, beginning 8 months (32 weeks) from drug initiation.
  Toxicity profile (CTCAE criteria)
Tolerability of drug | 8 months (32 weeks) from drug initiation
  Intra-patient, maximum tolerated dose
Safety of drug | 8 months (32 weeks) from drug initiation
  Toxicity profile (CTCAE criteria)
Clonal evolution on bitopertin | Annually for up to 3 years, beginning 8 months (32 weeks) from drug initiation
  Rates of clonal evolution as measured by karyotypic, histologic, and flow cytometric changes
Rate of overall survival | Ongoing for up to 3 years, beginning 8 months (32 weeks) from drug initiation
  Rate of overall survival according to clinical outcomes
Health-related quality of life (HRQL) | Annually for up to 3 years, beginning 8 months (32 weeks) from drug initiation
  Questionnaire-based inventory of HRQL

CONTACTS AND LOCATIONS:
Overall Officials: David J Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will generate data as specified by the clinical protocol, including patient characteristics/demographics and primary/secondary outcomes. To protect research participant identities, individual de-identified data points will be made available.@@@Sufficient data produced in the course of the project will be preserved. Sufficient data produced will also be shared except if limited by patient request (i.e., informed consent), federal or local laws and regulations (e.g., Health Insurance Portability and Accountability Act/HIPAA), or within the embargo period specified by the Cooperative Research and Development Agreement (CRADA) associated with this project (HL-CTCR-22-08002).@@@The project does not involve any data collection instruments that would limit accessibility or interpretation of the scientific data. To facilitate interpretation of the data, applicable protocol case report form templates, protocol, and data dictionaries, will be shared and associated with the relevant datasets.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available by the end of the protocol or at the time of associated publication, whichever comes first.
Access Criteria: BioData Catalyst is supported by NHLBI and access to data is controlled by the NHLBI Data Access Committee (DAC) utilizing the database of Genotypes and Phenotypes (dbGaP) permissions infrastructure. In order to access controlled-access data in BioData Catalyst, an investigator must have an approved Data Access Request (DAR) in dbGaP.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001528-H.html